CLINICAL TRIAL: NCT01573013
Title: Interactions of Lead Intoxication and Iron Deficiency in Morocco: The Effects of Iron Fortification With and Without NaEDTA on Lead Burden, Iron Status and Cognition in Children
Brief Title: Iron Fortification Trail Using NaFeEDTA in Iron Deficient Lead-exposed Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr. med, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: IZ70Z0_123902; IZ70Z0_123902 (Other Grant/Funding Number: The Swiss National Science Foundation (SNSF)/Project Nr. IZ70Z0_123902)
Record Dates: First submitted 2011-11-08; First posted 2012-04-06 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Iron Deficiency; Lead Poisoning
Keywords: iron deficiency; Lead poisoning; cognitive development; motor activity
MeSH Terms: conditions — Iron Deficiencies; Lead Poisoning; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NaFeEDTA treatment, biscuit (Active Comparator): Group receives 10 mg of Fe in form of NaFeEDTA per day. wheat flour based biscuit
  Interventions: Dietary Supplement: iron fortified biscuits
- EDTA treatment, biscuit (Active Comparator): Group receives Na2EDTA enriched biscuit
  Interventions: Dietary Supplement: iron fortified biscuits
- FeSO4 treatment, biscuit (Active Comparator): Group receives 10 mg of iron as FeSo4 per day for 8 months
  Interventions: Dietary Supplement: iron fortified biscuits
- control treatment, biscuit (Placebo Comparator): group receives a biscuit without additional iron
  Interventions: Dietary Supplement: iron fortified biscuits

INTERVENTIONS:
Dietary Supplement: iron fortified biscuits — 10 mg of iron per day for 8 months, either in the form of NaFeEDTA
  Arms: NaFeEDTA treatment, biscuit
Dietary Supplement: iron fortified biscuits — 10 mg of iron per day for 8 months, in the form of FeSo4
  Arms: FeSO4 treatment, biscuit
Dietary Supplement: iron fortified biscuits — EDTA fortified biscuit on a daily basis for 8 months
  Arms: EDTA treatment, biscuit
Dietary Supplement: iron fortified biscuits — control biscuit on a daily basis for 8 months
  Arms: control treatment, biscuit

SUMMARY:
In a cross-sectional study allotted by the ethical committee of the ETH Zurich, we are investigating the extent of anemia, iron deficiency and lead intoxication in young children. For this purpose an assessment of body lead burden and iron status was conducted in a cohort of individuals residing in areas of presumed high lead exposure. Associations between lead burden and iron status will be investigated in the near future (current status of the study).

In a follow-on intervention study, the effect of iron fortification with and without NaEDTA on blood lead levels in lead-exposed children will be evaluated; and the relative impact of these two strategies on child growth, motor and cognitive test performance will be compared.

This study will investigate the potential use of iron fortification to not only combat anemia but also reduce body lead burden in lead-exposed populations; it specifically investigates whether iron fortification with NaFeEDTA could have additional beneficial effects to iron alone.

DETAILED DESCRIPTION:
Introduction Coexisting chronic lead poisoning and iron deficiency anemia (IDA) are common in urban areas in developing regions, particularly in young children. In urban Morocco, anemia affects more than 1/3rd of schoolchildren and lead exposure is high. Lead poisoning and IDA both impair cognitive development and educability and may therefore have substantial health, social and economic costs on developing countries.

Iron status alters susceptibility to gastrointestinal lead exposure; absorption of lead is sharply increased in children with IDA. IDA upregulates the divalent metal transporter trans-port protein (DMT-1) and increases lead absorption. Thus, iron fortification to reduce IDA may also reduce lead absorption and be an effective strategy to accompany environmental lead abatement. The optimal iron compound for wheat flour is currently debated, and although elemental iron compounds are commonly used, they may be only poorly absorbed in the face of inhibitory compounds found in wheat flour.

A form of chelated iron, NaFeEDTA, is a promising iron fortificant that is recommended for wheat flour fortification. It is also a lead chelator. It may be superior to other iron fortificants in its ability to reduce body lead burden, due to:

1. its iron is highly bioavailable in the face of dietary inhibitors (such as phytic acid in wheat flour); and
2. potentially, its ability to chelate lead in the gut and bloodstream. Thus, it may be a good choice for fortification of wheat flour in Morocco, particularly in urban areas, to both reduce IDA and lower body lead.

Study aims and objectives:

1. Assessment of body lead burden and iron status in a cohort of individuals residing in areas of presumed high lead exposure. Investigation of associations between lead burden and iron status.
2. Comparison of effect of iron fortification with and without NaEDTA on body lead and iron status in lead-exposed children; and the relative impact on cognition.

Study hypotheses:

The prevalence of iron deficiency and elevated blood lead will be high in children in this region.

2) Body lead burden, as assessed by blood lead levels and urinary lead and delta-aminolevulinic acid (ALA), will be higher in individuals with poorer iron status.

3) Poor iron status will be associated with low intakes of bioavailable iron. 4) Greater severity of iron deficiency and/or higher body lead in children will predict poorer performance on cognitive and motor tests, and these conditions will interact to predict poorer performance.

Study design:

Our studies will be carried out in one of the four sub-economic areas, that were previously used in the baseline assessment in and near Marrakesh, Morocco (exact site still needs to be determined according to extend of lead contamination on the level of human population). Body lead burden and iron status will be determined, and associations between these examined using a cross-sectional design. For this purpose, blood and urine samples will be collected from two groups (preschool and school-aged children), residing in an area of high lead exposure.

Study design:

An 8-month intervention study in iron deficient, lead-exposed school children (n=500) will be designed to investigate whether iron fortification to reduce IDA may also reduce lead absorption and be an effective strategy to accompany environmental lead abatement.

For this purpose these children will be divided into four groups to receive a daily fortified baked snack containing either: 1) 66.4 mg NaFeEDTA ; 2) 52.2 mg Na2EDTA dehydrate; 3) 27.1 mg FeSO4 ; or 4) no fortificants.

ELIGIBILITY:
Inclusion Criteria:

* school and preschool children living in a lead-exposed environment with a high prevalence of iron deficiency

Exclusion Criteria:

* chronic or severe illnesses
* history of bleeding disorder

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 457 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
body lead burden | 8 months
  changes in blood lead levels over time of the intervention

SECONDARY OUTCOMES:
Iron status | 8 months
  changes in iron status (SF,Hb, TfR) before and after intervention
cognitive development | 8 months
  changes in cognitive development (using the K ABC II) before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof. Dr. med, Principal Investigator — Swiss Federal Institute of Technology (ETH)
Locations (1):
- Swiss Federal Institute of Technology (ETH), Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Bouhouch RR, El-Fadeli S, Andersson M, Aboussad A, Chabaa L, Zeder C, Kippler M, Baumgartner J, Sedki A, Zimmermann MB. Effects of wheat-flour biscuits fortified with iron and EDTA, alone and in combination, on blood lead concentration, iron status, and cognition in children: a double-blind randomized controlled trial. Am J Clin Nutr. 2016 Nov;104(5):1318-1326. doi: 10.3945/ajcn.115.129346. Epub 2016 Oct 12. PMID 27733396